CLINICAL TRIAL: NCT05862974
Title: A Randomized, Double-blind, Placebo-controlled, Dose-increasing Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Intravenous Infusion of LPM3480392 Injection in Healthy Subject
Brief Title: A Dose-escalation Study of LPM3480392 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY03014/CT-CHN-101
Record Dates: First submitted 2021-12-06; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- LPM3480392 X1mg (Experimental): 8 subjects will receive LPM3480392 X1mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X2mg (Experimental): 8 subjects will receive LPM3480392 X2 mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X3mg (Experimental): 8 subjects will receive LPM3480392 X3mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X4mg (Experimental): 8 subjects will receive LPM3480392 X4mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X5mg (Experimental): 8 subjects will receive LPM3480392 X5mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X6mg (Experimental): 8 subjects will receive LPM3480392 X6mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X7mg (Experimental): 8 subjects will receive LPM3480392 X7mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo
- LPM3480392 X8mg (Experimental): 8 subjects will receive LPM3480392 X8mg and 2 receive placebo
  Interventions: Drug: LPM3480392; Drug: Placebo

INTERVENTIONS:
Drug: LPM3480392 — Intravenous infusion of 30min duration
Drug: Placebo — Intravenous infusion of 30min duration

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-increasing Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single intravenous infusion of LPM3480392 injection in healthy subject

DETAILED DESCRIPTION:
A total of 80 healthy subjects will be allocated to 1 of 8 cohorts (cohort 1~8) in the study, each cohort including 10 subjects (8 subjects will receive investigational new drug (IND) product and 2 receive placebo). Each subject in fasted state will be randomly assigned to receive a single dose of LPM3480392 or placebo intravenously.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily signs the informed consent;
* Healthy male, aged 18-45 years (including boundary values);
* Body mass index (BMI) 19-26kg/m2 (including boundary value), weight ≥50kg;
* Subjects are willing to take contraceptive measures and promise not to donate sperm during the study period and within 90 days after administration;
* Willing to accept cold pain test, and the non-dominant hand can be soaked in ice water bath at 2℃ (± 0.2℃) for > 10s, < 120s.

Exclusion Criteria:

* Known history of allergy to any component of the investigational product or similar drugs, or allergic constitution [subjects with previous allergy to two or more foods or drugs];
* Past or present with any clinically significant disease or chronic disease of the respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, hematology, psychiatry, dermatology, orthostatic hypotension, etc.; or any disease that may interfere with the test results or interpretation of the results;
* Patients with Raynaud's syndrome;
* The skin wounds or skin diseases that may affect the cold pain test results; Sitting systolic blood pressure (SBP) < 90 mmHg, ≥ 140 mmHg or diastolic blood pressure (DBP) < 60 mmHg, ≥ 90 mmHg; subjects with heart rate < 60 beats/min, > 100 beats/min;
* QTc > 450 ms on electrocardiogram;
* Positive urine nicotine test;
* History of alcohol abuse within 3 months prior to Screening, defined as consumption of more than 14 units of alcohol per week (1 unit = 360 mL of beer, or 45 mL of spirits of 40% alcohol content, or 150 mL of wine), or a positive breath alcohol result;
* History of drug abuse or drug abuse or positive result of urine drug screening;
* Those who consume more than 100 g of xanthine-rich foods such as chocolate per day on average; those who consume more than 100 g of foods containing grapefruit and/or pomelo; those who consume more than 1000 mL of strong tea, coffee, cola and beverages containing caffeine and/or grapefruit ingredients.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Incidents of AE (including SAE) | from baseline to day8
  (including abnormal value of Vital signs,physical examination,laboratory tests,12-lead ECG)
DEQ | from baseline to day2
  Drug effect questionnaire,
OWS | from baseline to day3
  Opiate Withdrawal Scale

SECONDARY OUTCOMES:
AUC0-t | baseline and 48 hours after administration
  Pharmacokinetic index
AUC0-∞ | baseline and 48 hours after administration
  Pharmacokinetic index
Cmax | baseline and 48 hours after administration
  Pharmacokinetic index
Tmax | baseline and 48 hours after administration
  Pharmacokinetic index
T1/2 | baseline and 48 hours after administration
  Pharmacokinetic index
CL | baseline and 48 hours after administration
  Pharmacokinetic index
Vd | baseline and 48 hours after administration
  Pharmacokinetic index
MRT | baseline and 48 hours after administration
  Pharmacokinetic index
λz | baseline and 48 hours after administration
  Pharmacokinetic index
PD profile : Cold Pain Test | baseline and 8 hours after administration
  Pharmacodynamic index
PD profile : Pupillometry | baseline and 8 hours after administration
  Pharmacodynamic index

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hosipital zhejiang university school of medicine, Hangzhou, Zhejiang, China